CLINICAL TRIAL: NCT02354638
Title: Impact of Smoke Free Public Places (Smoke Free Cabs) on Cab Drivers in Mumbai, India
Brief Title: Impact of Smoke Free Public Places (Smoke Free Cabs) on Cab Drivers in Mumbai
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tata Memorial Hospital (Other Government)
Responsible Party: Principal Investigator, Gauravi Ashish Mishra, Associate Professor & Physician, Tata Memorial Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Screening
Other Study IDs: TMHPOCAB2015
Record Dates: First submitted 2014-12-11; First posted 2015-02-03 (Estimated); Last update posted 2018-04-30 (Actual); Status verified 2018-04

CONDITIONS: Compliance
Keywords: Perceptions; Education and evaluate post intervention KAP
MeSH Terms: conditions — Patient Compliance | interventions — Drug Therapy; Nicotine Replacement Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tobacco users: behavioural counseling (Experimental): The cab drivers using tobacco will be invited to participate in the tobacco cessation programme at the TCC and will receive three monthly follow-up for one year. Thus intervention will be in the form of behavioural therapy and pharmacotherapy (if required)
  Interventions: Behavioral: Tobacco users; Drug: Pharmacotherapy
- Non Users (No Intervention): The cab drivers who are not using tobacco in any form will not receive any type of intervention

INTERVENTIONS:
Behavioral: Tobacco users — Various tobacco cessation interventions in the form of one to one counseling, focus group discussions, role plays, games etc. will be used in the tobacco users.
  Arms: Tobacco users: behavioural counseling
Drug: Pharmacotherapy — Pharmacotherapy will also be prescribed as per the need assessment consisting of:
  Nicotine Chewing Gums:
  Dose: 2 mg/4 mg, 10-15 pieces per day with maximum dose of 24 pieces/day depending on cravings.Total Duration: 12 weeks Duration of treatment: Higher dose for 4-6 weeks, with weaning till 2-3 months
  Nicotine Transdermal patches:
  Dose: 7 mg/10 mg/14 mg/21 mg -for 24-hours use. Total Duration: 12 weeks Duration of treatment: Higher strength patch for 2 weeks and depending on cravings will be gradually decreased till 4 weeks
  Other Names: Nicotine replacement therapy
  Arms: Tobacco users: behavioural counseling

SUMMARY:
In addition to the passengers smoking inside the cab, the taxi drivers,are themselves addicted to smoking and/ or use of smokeless tobacco. Since tobacco is highly addictive, the cab drivers using tobacco need help in quitting. It is also necessary to raise the awareness of the cab drivers with respect to the hazards of tobacco and significance of the smoke free legislation.

It's been six years since the implementation of rules prohibiting smoking in public places and a re-look at the compliance to this regulation is necessary. The study will also help tobacco users to quit their habits. They will get screened for oral premalignant and malignant lesions.

Also, the cab drivers may pass on some effective messages regarding importance of keeping oneself away from tobacco, to the customers while commuting. In view of the above background, the current study is proposed to look at all these aspects.

The findings of the study will be certainly generating useful information with regards to lacunae in the existing system for appropriate implementation and for strengthening anti tobacco advocacy in our country.

DETAILED DESCRIPTION:
AIM and OBJECTIVES:

1. To study the Knowledge, Attitudes and Practices (KAP) regarding tobacco and smoke free public places among cab drivers ferrying customers near Tata Memorial Hospital
2. To study the impact of smoke free public places with specific reference to smoke free cabs (on various factors such as number of customers, customer practices, health status, self practices, compliance etc.)
3. To understand their attitude towards smoke free cabs.
4. To educate them regarding hazards of tobacco and the need for smoke free cabs.
5. To invite the cab drivers using tobacco to avail the Preventive Oncology screening facilities and Tobacco cessation clinic at the Tata Memorial Hospital
6. To evaluate the compliance for availing the services
7. To study the post-intervention KAP regarding tobacco and smoke free public places
8. To determine the rate of oral pre-cancers and tobacco cessation after one year follow-up.

Methodology:

Design: Single arm interventional study

Step 1: Around 400 cab drivers in Mumbai will be enrolled after explaining the programme and obtaining informed consent. They will be interviewed with the help of a well structured questionnaire to collect information about their Knowledge, Attitudes and Practices (KAP) regarding tobacco, their attitudes and experiences regarding smoke free public places with specific reference to smoke free cabs.

Step 2: The cab drivers will be given detailed health education regarding hazards of tobacco and the need for smoke free cabs. They will be invited to participate in oral cancer screening at the Preventive Oncology (PO) screening clinic.

Step 3: The cab drivers will be again interviewed with the help of a well structured questionnaire to collect information of their post-intervention KAP regarding tobacco and smoke free public places.

Step 4: The cab drivers using tobacco will be invited to participate in the tobacco cessation programme at the TCC and will receive three monthly follow-up for one year. Various tobacco cessation interventions in the form of one to one counseling, focus group discussions, role plays, games etc. will be used. In addition they will be engaged in conveying messages about tobacco control and refraining from tobacco habit, to the customers while commuting. This will also reinforce their own commitment towards tobacco cessation.

Variables to be estimated:

1. the change in the baseline KAP
2. the perceptions and attitude of cab drivers regarding implementation of smoke free cab policy.
3. the results of oral cancer screening in the form of oral pre-cancers and cancers detected
4. the success of tobacco cessation programme in the form of self reported quit rates at the end of one year
5. reactions of the commuters and their own perceptions towards the no tobacco messages conveyed to the customers while traveling

Data Analysis:

Data entry will be done in the Department of Preventive Oncology, Tata Memorial Hospital using SPSS version 18. Checks for consistency, data safety and analysis will be carried out at regular intervals. Both descriptive and inferential statistics will be generated for describing variables under the study objectives.

ELIGIBILITY:
Inclusion Criteria:

* 400 Cab drivers ferrying customers near Tata Memorial Hospital on a regular basis

Exclusion Criteria:

* Any Cab drivers outside the category as mentioned in the proposal

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2014-12; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Knowledge, Attitude & practice (change in the baseline KAP) | 30 months
  a) The

SECONDARY OUTCOMES:
Attitude regarding implementation of smoke free policy (perceptions and attitude of cab drivers) | 30 months
  b) The perceptions and attitude of cab drivers regarding implementation of smoke free cab policy.
Oral cancer detection by oral screening | 30 months
  c)The results of oral cancer screening in the form of oral pre-cancers and cancers detected
Quit rates (self reported quit rates) | 30 months
  d) The success of tobacco cessation programme in the form of self reported quit rates at the end of one year
Reactions towards no tobacco messages (Reactions of the commuters and their own perceptions) | 30 months
  e) Reactions of the commuters and their own perceptions towards the no tobacco messages conveyed to the customers while traveling

CONTACTS AND LOCATIONS:
Overall Officials: Gauravi A Mishra, Assoc Prof, Principal Investigator — Tata Memorial Hospital, Mumbai; Sharmila A Pimple, Professor, Principal Investigator — Tata Memorial Hospital, Mumbai
Locations (1):
- Gauravi A. Mishra, Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: Undecided